CLINICAL TRIAL: NCT06773078
Title: Validation of Urinary Biomarkers of Dietary Intake in Mexican Foods: a Randomize Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Responsible Party: Principal Investigator, Daniel Illescas Zárate, Doctorate in Science in Population Nutrition, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 5113
Record Dates: First submitted 2025-01-08; First posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Nutrition, Biomarkers of Intake, Urinary Biomarkers, Foodomics, Metabolom
Keywords: dietary assessment, nutrimetabolomics, avocado, corn tortilla, nopal, guava, mango, amaranth

STUDY DESIGN:
Intervention Model Description: Randomized controlled, open-label trial
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high intake group (Experimental): Intake of meals containing the foods of interest avocado, corn tortilla, nopal, guava, mango, amaranth in the breakfast.
  Interventions: Other: High intake group
- Average intake group (Experimental): Intake of meals containing the foods of interest avocado, corn tortilla, nopal, guava, mango, amaranth in the breakfast.
  Interventions: Other: Average intake group

INTERVENTIONS:
Other: High intake group — Intake of a breakfast containing the foods of interest avocado (80gr), corn tortilla (60 gr), nopal (200 gr), guava (108 gr), mango (100 gr), amaranth (14 gr).
  Arms: high intake group
Other: Average intake group — Intake of a breakfast containing the foods of interest avocado (40gr), corn tortilla (30 gr), nopal (100 gr), guava (54 gr), mango (50 gr), amaranth (7 gr).
  Arms: Average intake group

SUMMARY:
A randomized controlled open-label trial will be conducted in Mexico City, recruiting healthy participants who do not consume excessive alcohol or smoke. A selection visit will be conducted during which blood and urine samples will be collected, and assessments of diet, anthropometric measurements, and body composition will be performed.

DETAILED DESCRIPTION:
A randomized controlled open-label trial will be conducted in Mexico City, recruiting healthy participants who do not consume excessive alcohol or smoke. A selection visit will be conducted during which blood and urine samples will be collected, and assessments of diet, anthropometric measurements, and body composition will be performed.

Participants will be randomized into three groups for the intake of meals containing the foods of interest and control without these foods. After the meal consumption including foods of interest, a 24-hour urine sample will be collected by the participants. Urine and blood samples will be analyzed using using untargeted metabolomics in different platforms to determine biomarker concentrations.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Body mass index (BMI ) between 18.5 to 30 kg/m2
* Not having allergies to the study foods (ataulfo mango, nopal, guava, avocado, corn tortilla and amaranth).
* Without consumption of dietary supplements at the time of participating in the study.
* Blood chemistry within reference values (glucose <126 mg/dL, triglycerides <250 mg/dL, total cholesterol <250 mg/dL.

Exclusion Criteria:

* The exclusion criteria were participants with any other chronic disease diagnosed by any doctor.
* Were pregnant.
* Smoking habit durig the trial.
* Intake of alcoholic beverages during the trial.

Ages: 18 Years to 81 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Exploratory biomarkers of food intake | one day
  Mangiferin and pyrogallol for mango, peseitol, mannoheptulosa for avocado, and opuntiol for nopal.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No